CLINICAL TRIAL: NCT03690063
Title: Nice Human Immunodeficiency Virus (HIV) Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-DSP-01
Record Dates: First submitted 2018-09-17; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow up — Follow up of treatment, behavior, co-morbidity

SUMMARY:
Historically, the database on the HIV was organized within the framework of the medico-economic file of the human immunodeficiency (DMI-2), introduced jointly by the Direction of Hospitals (Mission AIDS) and the INSERM at the end of the 80s. Today this database is fed via the computerized medical record NADIS. Most part of the research works on the theme of the HIV take support on this database (DAD, EuroAIDS, Neuradapt).

ELIGIBILITY:
Inclusion Criteria:

* Enrol consecutive patients with a scheduled visit in the outpatient clinic (regardless of CD4 cell count and ART status).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients HIV innocents of any treatment and recently infected
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1996-01 (Actual); Primary Completion 1996-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
change of the clinico-biological signs of the patients | Each Year during 50 years
  change of the clinico-biological values form the start of the study, mesured every year, to the end of the study

SECONDARY OUTCOMES:
number of the various type of adverse events related by type of treatments | Each Year during 50 years
  Number of patients and laboratory data related to any events occurred such as : Death, Acute myocardial infarction , Ascites, Bone Mass Density , Diabetes mellitus, End Stage Renal Disease , Fibroscan stiffness , Bone fracture , Hepatic encephalopathy , Hepatorenal syndrome Invasive Cardiovascular Procedures , Kidney transplantation , Liver biopsy , Liver decompensation , Liver transplantation Non-AIDS defining malignancies , AIDS defining malignancies, Oesophageal variceal bleeding , Stroke

OTHER OUTCOMES:
number of the various type of co-morbidity | Each Year during 50 years
  Number of death, immediate cause of death, underlying conditions of death, ongoing risk factors in the year prior of the death, descripion of co-moirbidities (ongoing chronic conditions, prior cardiovascular diseases, history of depression, history of psychosis, liver diseases)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France